CLINICAL TRIAL: NCT00641550
Title: Effects of Physical Exercise During Pregnancy on the Maternal and Perinatal Outcomes: A Randomized Clinical Trial
Brief Title: Exercise and Pregnancy: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual da Paraiba (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Adriana Suely de Oliveira Melo, MD, MSc, Universidade Estadual da Paraiba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EXERC01
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Preeclampsia; Gestational Diabetes
Keywords: physical exercise; maternal complications; preterm labor; birthweight; Apgar scores
MeSH Terms: conditions — Pre-Eclampsia; Diabetes, Gestational; Motor Activity; Obstetric Labor, Premature; Birth Weight | interventions — Exercise; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Experimental): Pregnant women starting to practice physical exercise at 13 weeks(Walking moderate activity)
  Interventions: Other: Physical exercise
- 3 (Experimental): Pregnant women starting exercise at 20 weeks
  Interventions: Other: Physical exercise
- 1 (No Intervention): Pregnant women without exercise practice.

INTERVENTIONS:
Other: Physical exercise — Walking 3 times a week during 1 hours (moderate activity)
  Other Names: physical activity; physical exercise; walking
  Arms: 2; 3

SUMMARY:
The effects of physical exercise on pregnancy remain to be elucidated. A randomized controlled trial will be conducted to study the impact of exercise on maternal and perinatal outcomes. Our hypothesis is that physical exercise reduces preeclampsia incidence and improves birthweight when started early in pregnancy, with no impact on pregnancy duration, Apgar scores and neonatal complications.

DETAILED DESCRIPTION:
The study will include low risk pregnant women randomized to practice physical exercise beginning at 13 weeks, 20 weeks or no exercise group.

The objectives are:

1. To describe and compare biological and obstetrical variables.
2. To study doppler flow velocimetry indexes.
3. To determine the association between physical exercise and maternal complications: preeclampsia, preterm labor, gestational diabetes and weight gain in pregnancy.
4. To determine the association between physical exercise and perinatal outcomes: Apgar scores, birthweight, admission at intensive neonatal care unit, body composition and neonatal complications.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 13 weeks
* Single pregnancy
* Alive fetus
* No previous practice of physical activity

Exclusion Criteria:

* Smoking
* Chronic maternal diseases
* Placenta praevia
* History of preterm labor
* Bleeding

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 188 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Maternal outcome: preterm labor, weight gain, preeclampsia, gestational diabetes Perinatal outcome: birthweight, Apgar scores, body composition, admission at neonatal intensive care unit | nine months

SECONDARY OUTCOMES:
Doppler flow velocimetry indexes: pulsatility, resistance and A/B relation (uterine arteries, fetal middle cerebral artery and umbilical arteries) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Melania Amorim, PhD, Study Director — Instituto Materno Infantil Prof. Fernando Figueira
Locations (2):
- Brazil (2):
  - Universidade Estadual da Paraiba, Campina Grande, Paraíba
  - Universidade Estadual da Paraíba, Campina Grande, Paraíba

REFERENCES:
- [Derived] de Oliveria Melo AS, Silva JL, Tavares JS, Barros VO, Leite DF, Amorim MM. Effect of a physical exercise program during pregnancy on uteroplacental and fetal blood flow and fetal growth: a randomized controlled trial. Obstet Gynecol. 2012 Aug;120(2 Pt 1):302-10. doi: 10.1097/AOG.0b013e31825de592. PMID 22825089